CLINICAL TRIAL: NCT03641768
Title: Risk Prediction for Alzheimer Dementia With Brain Imaging and Genetics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not received
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00100030
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Alzheimer Dementia; Posttraumatic Stress Disorder; Traumatic Brain Injury
Keywords: Alzheimer Dementia; PTSD; MRI
MeSH Terms: conditions — Alzheimer Disease; Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Healthy volunteers (Active Comparator): Volunteers with no trauma history
  Interventions: Device: MRI; Device: PET; Device: 18F-Florbetapir; Device: Radioligand 18F-AV-1451
- Trauma only (Active Comparator): Volunteers that do not have PTSD but have had similar trauma to those with PTSD
  Interventions: Device: MRI; Device: PET; Device: 18F-Florbetapir; Device: Radioligand 18F-AV-1451
- PTSD only (Active Comparator): Volunteers with PTSD but no traumatic brain injury
  Interventions: Device: MRI; Device: PET; Device: 18F-Florbetapir; Device: Radioligand 18F-AV-1451
- PTSD and TBI (Active Comparator): Volunteers with PTSD and mild traumatic brain injury
  Interventions: Device: MRI; Device: PET; Device: 18F-Florbetapir; Device: Radioligand 18F-AV-1451

INTERVENTIONS:
Device: MRI — You will be asked to undergo a scan of your brain called an MRI. The MRI scan can measure the functioning of your brain.
Device: PET — You will be asked to undergo a scan of brain called a positron emission tomography (PET) scan. The PET scan is a test that uses radioactive glucose (sugar) and a computer to create images of how your brain is functioning. Abnormal cells in the body use glucose at a different rate than normal cells and this allows the scanner to create a detailed picture of how your body is working.
Device: 18F-Florbetapir — At the Duke University PET Center you will be in a quiet dimly lit space with only ambient room sound, with your eyes open and ears unplugged. Your safety will be monitored by a physician and nurse. 18F-florbetapir will be administered to you as a bolus injection through a peripheral vein followed by a flush and 10 minute continuous brain PET imaging will begin 50 minutes post-injection.
  Other Names: PET tracer for Amyloid-beta
Device: Radioligand 18F-AV-1451 — At the Duke University PET Center you will be in a quiet dimly lit space with only ambient room sound, with your eyes open and ears unplugged. Your safety will be monitored by a physician and nurse. 18F-florbetapir will be administered to you as a bolus injection through a peripheral vein followed by a flush and 10 minute continuous brain PET imaging will begin 50 minutes post-injection.
  Other Names: PET tracer for Tau protein

SUMMARY:
The purpose of this study is to learn about how trauma, posttraumatic stress disorder (PTSD), and mild traumatic brain injury that can occur during deployment affect the brain. The investigators also want to learn how PTSD and mild traumatic brain injury can affect the chance of developing Alzheimer disease later in life. The investigators will study this by using magnetic resonance imaging and positron emission tomography scans to obtain pictures of the brain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 65
* Previously enrolled in studies of OEF/OIF veterans by the same investigators
* Free of implanted metal objects or mental shards in eyes
* Fluent in English and capable of consenting

Exclusion Criteria:

* Axis I disorders other than Major Depressive Disorder or PTSD
* Current substance abuse or lifetime substance dependence (other than nicotine)
* High risk for suicide
* Claustrophobia
* Neurological disorders
* Learning disability or developmental delay
* Major medical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Cortical thickness as measured by MRI scans | Baseline
Beta amyloid plaques as measured by PET scans | Baseline
Tau proteins as measured by PET scans | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rajendra Morey, MD, Principal Investigator — Duke University
Locations (1):
- Durham VA, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No